CLINICAL TRIAL: NCT07031375
Title: Forest Bathing Programs in Families Receiving Early Intervention: A Feasibility Study
Brief Title: Forest Bathing Programs in Families Receiving Early Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202504055RINC
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Early Interventions
Keywords: Family-Centered; Green Care; Social Prescribing
MeSH Terms: interventions — Forest Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-Centered Forest Bathing Program (Experimental): Two-Day Family-Centered Forest Therapy Program
  Interventions: Behavioral: Social prescribing

INTERVENTIONS:
Behavioral: Social prescribing — This two-day family-centered forest therapy program incorporates the six core elements of Forest Therapy-plants, water, diet, psychology, climate, and exercise therapy-while integrating multi-sensory experiences and group interaction.
  Other Names: forest therapy

SUMMARY:
This study aims to develop and evaluate a two-day, one-night family-centered Forest Therapy program, exploring its feasibility and effectiveness on children's physical and psychological development as well as parental stress.

DETAILED DESCRIPTION:
The research plans to recruit 16 families, each consisting of one child aged 5 to 6 who is receiving early intervention services and both of their parents. The program incorporates the six core elements of Forest Therapy-plants, water, diet, psychology, climate, and exercise therapy-while integrating multi-sensory experiences and group interaction. Outcome evaluations will include physiological and psychological assessments, questionnaires, and interviews with both children and parents to examine pre- and post-intervention differences and gather feedback on the program.

ELIGIBILITY:
Inclusion Criteria:

1. child is currently between 5 years 0 months and 6 years 11 months of age and is receiving early intervention services.
2. child's language abilities (including communication and comprehension) and motor skills are at or above the developmental level of a typical three-year-old.
3. Family members (including two caregivers and the child receiving early intervention) are willing to fully participate in the two-day, one-night Forest Therapy program, including pre-test, post-test, and follow-up assessments.

Exclusion Criteria:

1. child has significant physical or motor impairments that affect mobility.
2. child is unable to understand instructions, which may hinder participation in activities.
3. Family members have allergies to the forest environment or other health risks that may be triggered by participation.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Actigraphy | 3 days before 2-day camp untile 3 days after camp
  Actigraphy is a non-invasive method of monitoring human rest/activity cycles.
Multidimensional Attention Test | Day 1 before the camp, day 2 immediately after the camp, 1 week after the camp
  The Multidimensional Attention Test (MAT) is a psychological assessment tool designed to evaluate different aspects of attention in children or adolescents.
Children's Motivation Questionnaire | Day-2 immediately after the camp
  Designed to evaluate children's motivation in engaging with tasks or activities

SECONDARY OUTCOMES:
Parent-Child Relationship Inventory | Day 1 before the camp, day 2 immediately after the camp, 1 week after the camp
  The Parent-Child Relationship Inventory (PCRI) assesses parents' attitudes toward parenting and their relationship with their child, covering support, involvement, communication, and discipline.
Parenting Stress Index-Four Edition short form | Day 1 before the camp, day 2 immediately after the camp, 1 week after the camp
  The Parenting Stress Index, Fourth Edition Short Form (PSI-4-SF) is a 36-item questionnaire designed to quickly assess parenting stress. It evaluates three core domains: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, helping identify stress levels that may affect parent-child relationships and guide intervention.
Satisfaction Questionnaire | Day 2 immediately after the camp
  To measure individuals' perceived satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Ni Wang, PhD, Principal Investigator — National Taiwan University, Department of Occupational Therapy
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No